CLINICAL TRIAL: NCT03158584
Title: Safety and Efficacy of Intrathecal Morphine in Children Undergoing Major Abdominal Surgeries, Dose-finding Clinical Study
Brief Title: Effect of Intrathecal Morphine in Children Undergoing Major Abdominal Surgeries,
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sahar Abdel Baky Mohamed, Assistant Professor of Anesthesia,Intensive care and Pain relief, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 343
Record Dates: First submitted 2017-05-14; First posted 2017-05-18 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2016-07

CONDITIONS: Major Abdominal Surgeries
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- morphine 2 μg/kg (Active Comparator): Children will receive intrathecal morphine 2 μg/kg in 2 ml volume normal saline.
  Interventions: Drug: Intrathecal Morphine
- morphine 5 μg/kg (Active Comparator): Children will receive intrathecal morphine 5 μg/kg in 2 ml volume normal saline.
  Interventions: Drug: Intrathecal Morphine
- morphine 10 μg/kg (Active Comparator): Children will receive intrathecal morphine 10 μg/kg in 2 ml volume normal saline.
  Interventions: Drug: Intrathecal Morphine

INTERVENTIONS:
Drug: Intrathecal Morphine — Intrathecal administration of Morphine in children undergoing major abdominal surgeries
  Other Names: morphine sulphate

SUMMARY:
safety and efficacy of intrathecal morphine in post operative pain relief in pediatric patients undergoing major abdominal cancer surgeries using different doses of intrathecal morphine (2 μg/kg , 5 μg/kg ,10 μg/kg).

DETAILED DESCRIPTION:
After obtaining approval of the local ethics committee of faculty of medicine, Assiut University , Assiut , Egypt , and parent's written informed consent, This randomized double -blinded prospective study conducted on ( 45 ) pediatric patients aged 3-12 years , weighting between 10-30 kg , and of American Society of Anesthesiologists (ASA) physical status I and II scheduled for major abdominal surgeries

ELIGIBILITY:
Inclusion Criteria

* weight between 10-30 kg ,
* American Society of Anesthesiologists (ASA) I - II
* major abdominal surgeries

Exclusion Criteria

* Children with sacral bone abnormalities
* spina bifida
* coagulopathy
* mental delay or retardation

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-07-01 (Estimated)

PRIMARY OUTCOMES:
visual analog scale | 24 hours postoperative .
  0- 10 in cm score range will be used to assess pain

SECONDARY OUTCOMES:
rams y sedation score | 24 hours
  0-4 score will be used

CONTACTS AND LOCATIONS:
Overall Officials: Sahar A Mohamed, MD, Principal Investigator — south egypt cancer instutite
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided